CLINICAL TRIAL: NCT04972110
Title: Phase 1b/2 Study of ATR InhibiTor RP-3500 and PARP Inhibitor Combinations in Patients With Molecularly Selected Cancers (ATTACC)
Brief Title: Study of RP-3500 (Camonsertib) With Niraparib or Olaparib in Advanced Solid Tumors
Acronym: ATTACC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to terminate study early therefore, the Phase 2 portion was not conducted
Sponsor: Repare Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP-3500-03
Record Dates: First submitted 2021-07-02; First posted 2021-07-22 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor, Adult
MeSH Terms: interventions — niraparib; olaparib

STUDY DESIGN:
Intervention Model Description: Dose Escalation, expansion and Phase 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase Ib Dose Escalation (Experimental): Multiple dose levels of RP-3500 (camonsertib) for oral administration in combination with niraparib and/or Multiple dose levels of RP-3500 (camonsertib) for oral administration in combination with olaparib
  Interventions: Drug: RP-3500 (camonsertib)
- Phase 2 Expansion Cohorts (Experimental): Expansion cohort with RP-3500 (camonsertib) + niraparib and/or Expansion cohort RP-3500 (camonsertib) + olaparib
  Interventions: Drug: RP-3500 (camonsertib)

INTERVENTIONS:
Drug: RP-3500 (camonsertib) — RP-3500 (camonsertib, ATR inhibitor) in combination with niraparib or olaparib (PARP inhibitors)
  Other Names: niraparib; olaparib

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of niraparib or olaparib in combination with RP-3500 (camonsertib), in patients with eligible advanced solid tumors, determine the maximum tolerated dose (MTD) of RP-3500 (camonsertib) in combination with niraparib or olaparib, examine pharmacokinetics (PK) and assess anti-tumor activity.

DETAILED DESCRIPTION:
This is a first-in-human Phase 1b/2, multi-center, open-label, dose-escalation and expansion study to:

* Evaluate the safety profile and MTD of RP-3500 (camonsertib) when administered orally in combination with niraparib or olaparib to establish the recommended Phase 2 dose and schedule.
* Characterize the PK profile of RP-3500 (camonsertib) in combination with niraparib or olaparib
* Assess anti-tumor activity associated with RP-3500 (camonsertib) in combination with niraparib or olaparib
* Examine biomarker responses and establish a correlation with RP-3500 (camonsertib) treatment in combination with niraparib or olaparib.

After the RP2D and schedule is determined, expansion cohort(s) for RP-3500 (camonsertib) in combination with niraparib or olaparib will be enrolled to study the anti-tumor effect, and further examine the safety, PK, and pharmacodynamic (PD).

Sponsor decided to terminate study early therefore, the Phase 2 expansion was not conducted

ELIGIBILITY:
Inclusion Criteria:

* Male or female and ≥18 years-of-age at the time of signature of the informed consent
* Confirmed advanced solid tumors resistant or refractory to standard treatment
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Evaluable disease as per RECIST v1.1
* Next generation sequencing (NGS) report obtained in CLIA-certified or equivalent laboratory demonstrating eligible tumor biomarkers.
* Submission of available tumor tissue or willingness to have a biopsy performed if safe and feasible
* Acceptable hematologic and organ function at screening
* Negative pregnancy test for women of childbearing potential at Screening and prior to first study drug.
* Ability to swallow and retain oral medications.

Exclusion Criteria:

* Prior therapy with an ATR or DNA-dependent protein kinase (DNA-PK) inhibitor.
* Chemotherapy, small molecule anticancer or biologic anticancer therapy given within 10 days or 5 half-lives (whichever is longer), prior to first dose of study drug.
* Use of radiotherapy (except for palliative reasons) within 7 days prior to first dose of study drug.
* History or current condition, therapy, or laboratory abnormality that might confound the study results, or interfere with the patient's participation for the full duration of the study treatment.
* No other anticancer therapy is to be permitted while the patient is receiving study treatment.
* Major surgery ≤28 days or minor surgical procedures ≤7 days prior to first study treatment dose.
* Uncontrolled, symptomatic brain metastases.
* Uncontrolled high blood pressure
* History of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) diagnosis
* Presence of other known active invasive cancers.
* Pregnant or breastfeeding women.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the study protocol and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Participating Site #1018, Phoenix, Arizona
  - Participating Site #1025, San Francisco, California
  - Participating Site #1028, Aurora, Colorado
  - Participating Site #1012, New Haven, Connecticut
  - Participating Site #1017, Jacksonville, Florida
  - Participating Site #1009, Baltimore, Maryland
  - Participating Site #1015, Ann Arbor, Michigan
  - Participating Site # 1016, Rochester, Minnesota
  - Participating Site #1026, New York, New York
  - Participating Site # 1008, New York, New York
  - Participating Site #1029, Eugene, Oregon
  - Participating Site # 1001, Houston, Texas
  - Participating Site # 1013, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silverman IM, Schonhoft JD, Herzberg B, Yablonovitch A, Lagow E, Fiaux PC, Safabakhsh P, Sethuraman S, Ulanet D, Yang J, Kim I, Basciano P, Cecchini M, Lee E, Lheureux S, Fontana E, Carneiro BA, Reis-Filho JS, Yap TA, Zinda M, Rosen EY, Rimkunas V. Genomic and Epigenomic ctDNA Profiling in Liquid Biopsies from Heavily Pretreated Patients with DNA Damage Response-Deficient Tumors. Clin Cancer Res. 2025 Oct 1;31(19):4136-4149. doi: 10.1158/1078-0432.CCR-25-1248. PMID 40705098

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: 50mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly: 50 mg RP-3500 (camonsertib) taken QD (once a day) orally in combination with 100 mg niraparib taken QD orally, same day on a 3 days on and 4 days off schedule for 3 weeks (21 day cycle)
- Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly: 80 mg RP-3500 (camonsertib) taken QD orally in combination with 100 mg niraparib taken QD orally, same day on a 2 days on and 5 days off schedule for 3 weeks (21 day cycle)
- Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly: 80 mg RP-3500 (camonsertib) taken QD orally in combination with 100 mg niraparib taken QD orally, same day on a 3 days on and 4 days off schedule for 3 weeks (21 day cycle)
- Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, 2 weeks on/1 week off: 80 mg RP-3500 (camonsertib) taken QD orally in combination with 100 mg niraparib taken QD orally, same day on a 2 days on and 5 days off schedule for 2 weeks on and 1 week off (21 day cycle)
- Arm 1: 70mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly: 70 mg RP-3500 (camonsertib) taken QD orally in combination with 100 mg niraparib taken QD orally, same day on a 2 days on and 5 days off schedule for 3 weeks (21 day cycle)
- Arm 2: 50mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly: 50 mg RP-3500 (camonsertib) taken QD orally in combination with 150 mg olaparib taken BID (twice a day) orally, same day on a 3 days on and 4 days off schedule for 3 weeks (21 day cycle)
- Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 3d on/4d off, weekly: 50 mg RP-3500 (camonsertib) taken QD orally in combination with 100 mg olaparib taken BID orally, same day on a 3 days on and 4 days off schedule for 3 weeks (21 day cycle)
- Arm 2: 50mg QD camonsertib + 200 mg QD olaparib, 3d on/4 d off, weekly: 50 mg RP-3500 (camonsertib) taken QD orally in combination with 200 mg olaparib taken QD orally, same day on a 3 days on and 4 days off schedule for 3 weeks (21 day cycle)
- Arm 2: 80mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly: 80 mg RP-3500 (camonsertib) taken QD orally in combination with 150 mg olaparib taken BID orally, same day on a 3 days on and 4 days off schedule for 3 weeks (21 day cycle)
- Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, weekly: 50 mg RP-3500 (camonsertib) taken QD orally in combination with 100 mg olaparib taken BID orally, same day on a 2 days on and 5 days off schedule for 3 weeks (21 day cycle)
- Arm 2: 80mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, 2w on/1w off: 80 mg RP-3500 (camonsertib) taken QD orally in combination with 100 mg olaparib taken BID orally, same day on a 2 days on and 5 days off schedule for 2 weeks on and 1 week off (21 day cycle)
Period: Overall Study
Arm/Group | Arm 1: 50mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, 2 weeks on/1 week off | Arm 1: 70mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 200 mg QD olaparib, 3d on/4 d off, weekly | Arm 2: 80mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, weekly | Arm 2: 80mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, 2w on/1w off
Started | 9 | 24 | 3 | 23 | 8 | 7 | 19 | 5 | 3 | 26 | 29
Completed | 1 | 4 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Not Completed | 8 | 20 | 2 | 23 | 8 | 7 | 18 | 4 | 2 | 26 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: 50mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, 2 weeks on/1 week off | Arm 1: 70mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 200 mg QD olaparib, 3d on/4 d off, weekly | Arm 2: 80mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, weekly | Arm 2: 80mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, 2w on/1w off | Total
Number analyzed (Participants) | 9 | 24 | 3 | 23 | 8 | 7 | 19 | 5 | 3 | 26 | 29 | 156
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 60.9 (13.51) | 61.7 (7.70) | 61.7 (15.18) | 56.4 (9.01) | 63.1 (12.14) | 53.1 (14.24) | 56.8 (14.60) | 59.8 (12.40) | 59.3 (21.08) | 58.8 (13.38) | 59.2 (13.73) | 58.9 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 20 | 2 | 19 | 8 | 3 | 12 | 2 | 1 | 15 | 16 | 104
  Male | 3 | 4 | 1 | 4 | 0 | 4 | 7 | 3 | 2 | 11 | 13 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 11
  Not Hispanic or Latino | 9 | 22 | 3 | 18 | 8 | 6 | 18 | 5 | 3 | 23 | 26 | 141
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Determine the Safety and Tolerability of Niraparib or Olaparib in Combination With RP-3500 in Patients With Molecularly Selected Solid Tumors
Description: Treatment Related Treatment-Emergent Adverse Events (TRAE) with ≥3 CTCAE Grade
Time Frame: Start of treatment to 30 days post last dose, up to 23.7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 50mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, 2 weeks on/1 week off | Arm 1: 70mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 200 mg QD olaparib, 3d on/4 d off, weekly | Arm 2: 80mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, weekly | Arm 2: 80mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, 2w on/1w off
Number analyzed (Participants) | 9 | 24 | 3 | 23 | 8 | 7 | 19 | 5 | 3 | 26 | 29
Participants | 8 | 20 | 3 | 12 | 7 | 6 | 16 | 5 | 3 | 16 | 23

2. Primary Outcome: Define the Recommended Phase 2 Dose (RP2D) of RP-3500 in Combination With Niraparib or Olaparib in Patients With Molecularly Selected Solid Tumors
Description: Frequency of DLTs during the DLT observation period
Time Frame: During 21 days (one cycle) from the initiation of the study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 50mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, 2 weeks on/1 week off | Arm 1: 70mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 200 mg QD olaparib, 3d on/4 d off, weekly | Arm 2: 80mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, weekly | Arm 2: 80mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, 2w on/1w off
Number analyzed (Participants) | 8 | 22 | 3 | 22 | 8 | 6 | 17 | 4 | 3 | 26 | 27
Participants | 1 | 1 | 3 | 1 | 1 | 3 | 6 | 1 | 2 | 0 | 3

ADVERSE EVENTS:
Time Frame: Start of treatment to 30 days post lase dose, up to 34.7 months for Serious adverse events; Start of treatment to 30 days post last dose, up to 23.7 months for other adverse events
Groups:
- Arm 1: 70mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly: 70 mg RP-3500 (camonsertib) taken QD orally in combination with 100 mg niraparib taken QD orally, same day on a 2 days on and 5 days off schedule for 3 weeks (21 day cycle)
Arm/Group | Arm 1: 50mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, 2 weeks on/1 week off | Arm 1: 70mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly | Arm 2: 50mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 200 mg QD olaparib, 3d on/4 d off, weekly | Arm 2: 80mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, weekly | Arm 2: 80mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, 2w on/1w off
All-Cause Mortality (participants affected / at risk) | 3/9 | 10/24 | 0/3 | 8/23 | 1/8 | 4/7 | 10/19 | 1/5 | 1/3 | 6/26 | 5/29
Serious Adverse Events (participants affected / at risk) | 4/9 | 8/24 | 2/3 | 7/23 | 3/8 | 1/7 | 11/19 | 2/5 | 1/3 | 8/26 | 8/29
Other Adverse Events (participants affected / at risk) | 9/9 | 24/24 | 3/3 | 23/23 | 8/8 | 7/7 | 19/19 | 5/5 | 3/3 | 26/26 | 27/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: 50mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly (N=9) | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly (N=24) | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly (N=3) | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, 2 weeks on/1 week off (N=23) | Arm 1: 70mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly (N=8) | Arm 2: 50mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly (N=7) | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 3d on/4d off, weekly (N=19) | Arm 2: 50mg QD camonsertib + 200 mg QD olaparib, 3d on/4 d off, weekly (N=5) | Arm 2: 80mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly (N=3) | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, weekly (N=26) | Arm 2: 80mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, 2w on/1w off (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Neutrophil count decreased/ Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Platelet count decreased/ Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders and administration site conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: 50mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly (N=9) | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly (N=24) | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 3d on/4d off, weekly (N=3) | Arm 1: 80mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, 2 weeks on/1 week off (N=23) | Arm 1: 70mg QD camonsertib + 100mg QD niraparib, 2d on/5d off, weekly (N=8) | Arm 2: 50mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly (N=7) | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 3d on/4d off, weekly (N=19) | Arm 2: 50mg QD camonsertib + 200 mg QD olaparib, 3d on/4 d off, weekly (N=5) | Arm 2: 80mg QD camonsertib + 150mg BID olaparib, 3d on/4d off, weekly (N=3) | Arm 2: 50mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, weekly (N=26) | Arm 2: 80mg QD camonsertib + 100mg BID olaparib, 2d on/5d off, 2w on/1w off (N=29)
Anaemia (Blood and lymphatic system disorders) | 8 | 20 | 3 | 15 | 6 | 6 | 17 | 4 | 3 | 24 | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 4 | 0 | 2 | 0 | 2 | 1 | 2 | 0 | 2 | 4
Neutrophil count decreased/ Neutropenia (Blood and lymphatic system disorders) | 4 | 15 | 3 | 5 | 1 | 2 | 14 | 3 | 3 | 13 | 21
Platelet count decreased/ Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 10 | 3 | 3 | 0 | 4 | 7 | 2 | 1 | 5 | 11
WBC count decreased/ Leukopenia (Blood and lymphatic system disorders) | 3 | 8 | 1 | 1 | 0 | 1 | 10 | 3 | 1 | 8 | 10
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac discomfort (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 4 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 1 | 3 | 1 | 0 | 2 | 2 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 0 | 7 | 2 | 0 | 1 | 1 | 1 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 10 | 1 | 5 | 1 | 1 | 2 | 1 | 1 | 5 | 6
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 0 | 5 | 2 | 2 | 3 | 0 | 0 | 6 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 9 | 0 | 11 | 5 | 0 | 5 | 2 | 2 | 7 | 12
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 1 | 0 | 3 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 8 | 1 | 11 | 2 | 2 | 2 | 2 | 1 | 4 | 5
Asthenia (General disorders and administration site conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Axillary pain (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders and administration site conditions) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crying (General disorders and administration site conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deformity (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Early satiety (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders and administration site conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders and administration site conditions) | 4 | 17 | 2 | 9 | 3 | 2 | 7 | 3 | 2 | 9 | 10
Influenza like illness (General disorders and administration site conditions) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Localised oedema (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malaise (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2
Mucosal inflammation (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders and administration site conditions) | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Oedema peripheral (General disorders and administration site conditions) | 2 | 3 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 1 | 4
Pain (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders and administration site conditions) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders and administration site conditions) | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 2 | 1
Suprapubic pain (General disorders and administration site conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (General disorders and administration site conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders and administration site conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 5 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ludwig angina (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 3
Urinary tract infection (Infections and infestations) | 2 | 3 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urostomy complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 2 | 2 | 2 | 0 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 4 | 4
Blood albumin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 3 | 3
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Blood chloride decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nitrite urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroxine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Weight decreased (Investigations) | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 2 | 2 | 2 | 0 | 4 | 3 | 1 | 4 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 4 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 7 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 4 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 6 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aura (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 4 | 2 | 0 | 3 | 0 | 1 | 2 | 4
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 7 | 0 | 6 | 1 | 2 | 3 | 1 | 1 | 4 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 5 | 0 | 4 | 1 | 0 | 1 | 0 | 1 | 2 | 4
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penile discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 2 | 1 | 1 | 4 | 0 | 2 | 0 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 2 | 3 | 3 | 2 | 3 | 0 | 2 | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early. And phase 2 portion of the study was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT04972110/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT04972110/SAP_001.pdf